CLINICAL TRIAL: NCT05177783
Title: Contraception Decision Aid Use and Patient Outcomes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Texas Christian University (Other)
Responsible Party: Principal Investigator, Sarah Hill, Professor, Texas Christian University
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Supportive Care
Other Study IDs: TCU020519781
Record Dates: First submitted 2021-12-10; First posted 2022-01-05 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Contraceptive Usage
MeSH Terms: conditions — Contraception Behavior

STUDY DESIGN:
Intervention Model Description: Parallel
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants will be condition-blind (i.e., they will not be told whether the health application they use is the "treatment" or "control" application). Assignment to treatment arms will be randomized using Qualtrics Experimental Software and treatment assignment group will remain masked to the investigator and those in charge of data analysis until after data analysis is complete.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tuune (Experimental): Participants complete the Tuune contraceptive decision aid health questionnaire.
  Interventions: Behavioral: Tuune health questionnaire
- Control (Active Comparator): Participants complete a standard physician intake health questionnaire.
  Interventions: Behavioral: Control health questionnaire

INTERVENTIONS:
Behavioral: Tuune health questionnaire — Participants complete the Tuune contraceptive decision aid health questionnaire.
  Arms: Tuune
Behavioral: Control health questionnaire — Participants complete a standard physician intake health questionnaire.
  Arms: Control

SUMMARY:
The purpose of this study is to assess the impact of a contraception decision aid mobile application on: (a) decisional conflict, (b) reproductive health self-efficacy, (c) contraceptive and reproductive health literacy, and (d) contraceptive use intentions.

DETAILED DESCRIPTION:
After being informed about the study and the potential risks, all participants giving written informed consent will be randomly assigned in a double-blind manner (participant and investigator) in a 1:1 ratio to complete an interactive contraception decision aid health questionnaire (Tuune) or a standard medical questionnaire (Control). After, all participants will be asked questions assessing: (a) decisional conflict, (b) reproductive health self-efficacy, (c) contraceptive and reproductive health literacy, and (d) contraceptive use intentions.

ELIGIBILITY:
Inclusion Criteria:

* Females 18 to 34 years of age who enroll to participate in the study, which will take place on the campus of Texas Christian University.

Exclusion Criteria:

* Women who are currently pregnant or breastfeeding.
* Women who wish to become pregnant within the next 12 months.

Ages: 18 Years to 34 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 500 (Estimated)
Dates: Start 2022-01-15 (Actual); Primary Completion 2022-05-30 (Estimated); Study Completion 2022-08-30 (Estimated)

PRIMARY OUTCOMES:
Decisional Conflict | Immediately upon completion of the assigned health questionnaire.
  Decisional conflict about contraceptive use will be measured using a modified version of the "Traditional Decisional Conflict Scale" to assess decisional conflict about birth control use. The modified version of this scale is a 13-item measure utilizing a 1-7 rating scale (1 = strongly disagree | 7 = strongly agree) asking participants about their decisional conflict with respect to birth control. Higher scores on this scale indicate less decisional conflict about birth control use.
  A full list of items can be viewed on the Open Science Framework, here: https://osf.io/t4sq2/
  References:
  O'Connor AM (1995). Validation of a decisional conflict scale. Medical Decision Making, 15(1), 25-30. doi: 10.1177/0272989X9501500105.
Reproductive Health Self-Efficacy | Immediately upon completion of the assigned health questionnaire.
  Reproductive health self-efficacy will be measured using a modified version of the "Menstrual Attitudes Questionnaire". The modified version is a 9-item measure utilizing a 1-7 rating scale (1 = strongly disagree | 7 = strongly agree) asking participants about their menstrual cycle and hormonal self-efficacy. Higher scores indicate lower reproductive health self-efficacy.
  A full list of items can be viewed on the Open Science Framework, here: https://osf.io/t4sq2/
  References:
  Brooks-Gunn, J., & Ruble, D. N. (1980). The Menstrual Attitude Questionnaire. Psychosomatic Medicine, 42(5), 503-512. https://doi.org/10.1097/00006842-198009000-00005
Reproductive Health and Contraceptive Knowledge | Immediately upon completion of the assigned health questionnaire.
  Reproductive health and contraceptive knowledge will be measured using the following 6-item, 1-7 rating scale (1 = strongly disagree | 7 = strongly agree). Higher scores indicate greater reproductive health and contraceptive knowledge.
  A full list of items can be viewed on the Open Science Framework, here: https://osf.io/t4sq2/
Contraceptive Use Intentions | Immediately upon completion of the assigned health questionnaire.
  Contraceptive use intentions will be measured by asking participants to rate their likelihood of using hormonal birth control in the next week, month, and year. Each question will be measured on a 1-7 scale (1 = extremely unlikely to use | 7 = extremely likely to use). Higher scores indicate higher use intentions.
  A full list of items can be viewed on the Open Science Framework, here: https://osf.io/t4sq2/

SECONDARY OUTCOMES:
Patient Satisfaction | Immediately upon completion of the primary measures.
  Patient satisfaction with the health questionnaire will be measured using an intervention-tailored version of the "Clinical Use Satisfaction Scale". The modified version is a 14-item measure utilizing two 1-7 rating scales. Items 1 - 12 use the following rating scale: 1 = strongly disagree | 7 = strongly agree. Items 13 - 14 use the scale: 1 = very unlikely | 7 = very likely. Higher scores indicate greater satisfaction with the health questionnaire.
  A full list of items can be viewed on the Open Science Framework, here: https://osf.io/t4sq2/
  References:
  Zimmerman, M., Gazarian, D., Multach, M., Attiullah, N., Benoff, T., Boerescu, D. A., ... & Holst, C. G. (2017). A clinically useful self-report measure of psychiatric patients' satisfaction with the initial evaluation. Psychiatry research, 252, 38-44.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Hill, PhD, Principal Investigator — Texas Christian University
Locations (1):
- Texas Christian University, Fort Worth, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] O'Connor AM. Validation of a decisional conflict scale. Med Decis Making. 1995 Jan-Mar;15(1):25-30. doi: 10.1177/0272989X9501500105. PMID 7898294
- [Background] Brooks-Gunn J, Ruble DN. The menstrual attitude questionnaire. Psychosom Med. 1980 Sep;42(5):503-12. doi: 10.1097/00006842-198009000-00005. PMID 7465737
- [Background] Zimmerman M, Gazarian D, Multach M, Attiullah N, Benoff T, Boerescu DA, Friedman MA, Mehring LB, Moon S, Patel S, Holst CG. A clinically useful self-report measure of psychiatric patients' satisfaction with the initial evaluation. Psychiatry Res. 2017 Jun;252:38-44. doi: 10.1016/j.psychres.2017.02.036. Epub 2017 Feb 20. PMID 28242516
- [Derived] Espinosa M, Butler SA, Mengelkoch S, Prieto LJ, Russell E, Ramshaw C, Rose-Reneau Z, Remondino M, Nahavandi S, Hill SE. The Impact of a Digital Contraceptive Decision Aid on User Outcomes: Results of an Experimental, Clinical Trial. Ann Behav Med. 2024 Jun 18;58(7):463-473. doi: 10.1093/abm/kaae024. PMID 38828482